CLINICAL TRIAL: NCT06358222
Title: Predicting NSCLC Lymph Node Metastasis: Integrating ctDNA Mutation/ Methylation Profiling With PET-CT Scan: The LUNon-invasive Study
Brief Title: Predicting Non-small Cell Lung Cancer (NSCLC) Lymph Node Metastasis: Integrating Circulating Tumor DNA (ctDNA) Mutation/ Methylation Profiling With Positron Emission Tomography-computed Tomography (PET-CT) Scan
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Feng Yao, Professor, Shanghai Chest Hospital
Other Study IDs: LUNon-invasive
Record Dates: First submitted 2024-03-28; First posted 2024-04-10 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Carcinoma; Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; ctDNA; PET-CT; methylation; lymph node metastasis
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Lymphatic Metastasis | interventions — Methylation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Blood ctDNA + methylation + PET-CT vs Postoperative pathology
  Interventions: Procedure: Blood ctDNA + methylation + PET-CT and Postoperative pathology
- MRD+ methylation (or combined with PET-CT) vs Invasive mediastinoscopy /EBUS-TBNA
  Interventions: Procedure: MRD+ methylation (or combined with PET-CT) and Invasive mediastinoscopy /EBUS-TBNA
- Lymph Node dissection vs no lymph node dissection
  Interventions: Procedure: Intraoperative lymph node dissection

INTERVENTIONS:
Procedure: Blood ctDNA + methylation + PET-CT and Postoperative pathology — A highly sensitive tumor-naïve MRD panel of ctDNA will be employed to detect preoperative blood. Some patients will undergo methylation profiling to prospectively establish LNMs-specific ctDNA methylation signatures.
  Groups: Blood ctDNA + methylation + PET-CT vs Postoperative pathology
Procedure: MRD+ methylation (or combined with PET-CT) and Invasive mediastinoscopy /EBUS-TBNA — A certain number (depending on the Results of Stage 1) of patients requiring invasive mediastinoscopy or EBUS-TBNA, based on the clinical guidelines, will be included for blood ctDNA mutation/methylation profile (or combined PET-CT), and the detection rate of LNMs will be assessed in patients with negative preoperative blood ctDNA mutation/methylation (or combined PET-CT). The accuracy of predicting LNMs will be compared with that of patients with negative or positive preoperative blood ctDNA mutation/methylation (or combined PET-CT).
  Groups: MRD+ methylation (or combined with PET-CT) vs Invasive mediastinoscopy /EBUS-TBNA
Procedure: Intraoperative lymph node dissection — For patients with negative preoperative blood negative testing (ctDNA mutation/methylation profiles alone or in combination with PET-CT), systematic lymph node sampling/dissection and no lymph node dissection will be grouped and compared. Regular follow-up is performed to investigate the impact on long-term MRD negative duration and prognosis.
  Groups: Lymph Node dissection vs no lymph node dissection

SUMMARY:
This is a single center, prospective and observational study conducted in three stages to predict the NSCLC lymph node metastasis based on ctDNA/specific methylation molecular features combined with PET-CT imaging features and intervention study.

DETAILED DESCRIPTION:
This is a prospective study conducted in three stages. The volume of blood drawn will be 30 mL each time.

Stage 1: We will enroll 200 patients diagnosed with stage I-IIIB NSCLC who are scheduled for lobectomy and systematic lymph node dissection. The prediction of lymph node metastasis will be based on preoperative blood ctDNA mutation and methylation profiling. Specifically, during this stage, we will prospectively establish ctDNA methylation signatures specifically associated with LNMs in NSCLC. These molecular profiles will be combined with PET-CT imaging. Postoperative pathological results will serve as the reference standard for comparison.

Stage 2: A certain number (depending on the Results of Stage 1) of patients requiring invasive mediastinoscopy or EBUS-TBNA, based on the clinical guidelines, will be included for blood ctDNA mutation/methylation profile (or combined PET-CT), and the detection rate of LNMs will be assessed in patients with negative preoperative blood ctDNA mutation/methylation (or combined PET-CT). The accuracy of predicting LNMs will be compared with that of patients with negative or positive preoperative blood ctDNA mutation/methylation (or combined PET-CT).

Stage 3: For patients with negative preoperative blood negative testing (ctDNA mutation/methylation profiles alone or in combination with PET-CT), systematic lymph node sampling/dissection and no lymph node dissection will be grouped and compared. Regular follow-up is performed to investigate the impact on long-term MRD negative duration and prognosis. The primary outcomes: postoperative MRD negative duration and progression-free survival (PFS); The second outcomes: Overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to study initiation.
2. Age between 18 and 75 years.
3. Preoperative clinical evaluation indicating non-small cell lung cancer (NSCLC) stage I-IIIB (without initial treatment sought).
4. Newly treated patients who have consented to undergo surgery.
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0-1.

Exclusion Criteria:

1. Non-small cell lung cancer (NSCLC) histopathologically determined to be other than stage I-IIIB following surgical evaluation.
2. Presence of other active malignant tumor diseases.
3. Evidence of any serious or uncontrolled systemic illness, including uncontrolled hypertension and active bleeding, as assessed by the investigator, which may contribute to reluctance to participate in the trial or decrease adherence to the study regimen. Additionally, active infectious diseases such as hepatitis B, hepatitis C, and human immunodeficiency virus (HIV) infection are grounds for exclusion.
4. History of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis requiring steroid therapy, or any indication of clinically active ILD.
5. Patients considered by the investigator to be unable to comply with the study protocol, restrictions, and requirements, or those facing circumstances at the investigator's discretion that would impede their participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This program will be conducted in three stages. Stage 1: We will enroll 200 patients diagnosed with stage I-IIIB NSCLC who are scheduled for lobectomy and systematic lymph node dissection.
  Stage 2: A certain number (depending on the Results of Stage 1) of patients requiring invasive mediastinoscopy or EBUS-TBNA, based on the clinical guidelines, will be included for blood ctDNA mutation/methylation profile (or combined PET-CT), and the detection rate of LNMs will be assessed in patients with negative preoperative blood ctDNA mutation/methylation (or combined PET-CT).
  Stage 3: For patients with negative preoperative blood negative testing (ctDNA mutation/methylation profiles alone or in combination with PET-CT), systematic lymph node sampling/dissection and no lymph node dissection will be grouped and compared.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Negative prediction value (NPV) of lymph node metastasis rates | one day for each patient
  The primary endpoint will be the negative prediction value (NPV) of LNM rates between groups using preoperative blood ctDNA/methylation alone or in combination with PET-CT. LNMs-specific ctDNA methylation signatures will be developed and the sensitivity and specificity of ctDNA mutation/methylation profiles alone or when combined with PET-CT scans for predicting LNMs will be assessed. Postoperative pathological results will serve as the reference standard for comparison.
Disease-free survival (DFS) | Until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  DFS is defined as the time from surgical resection to tumor recurrence or death due to tumor progression. DFS will be compared between the ctDNA-positive group and the ctDNA-negative group. DFS will be assessed in stage 3.
ctDNA-free interval (CFI) | Until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years.
  CFI is defined as the duration between a patient's transition from ctDNA negative to ctDNA positive status.

SECONDARY OUTCOMES:
Overall Survival (OS) | Until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
  OS is defined as the time between the start of the patient's surgical resection and any documented death from any cause. OS will be compared between ctDNA-positive and ctDNA-negative groups. OS will be assessed in stage 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbosh C, Birkbak NJ, Wilson GA, Jamal-Hanjani M, Constantin T, Salari R, Le Quesne J, Moore DA, Veeriah S, Rosenthal R, Marafioti T, Kirkizlar E, Watkins TBK, McGranahan N, Ward S, Martinson L, Riley J, Fraioli F, Al Bakir M, Gronroos E, Zambrana F, Endozo R, Bi WL, Fennessy FM, Sponer N, Johnson D, Laycock J, Shafi S, Czyzewska-Khan J, Rowan A, Chambers T, Matthews N, Turajlic S, Hiley C, Lee SM, Forster MD, Ahmad T, Falzon M, Borg E, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Hafez D, Naik A, Ganguly A, Kareht S, Shah R, Joseph L, Marie Quinn A, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Oukrif D, Akarca AU, Hartley JA, Lowe HL, Lock S, Iles N, Bell H, Ngai Y, Elgar G, Szallasi Z, Schwarz RF, Herrero J, Stewart A, Quezada SA, Peggs KS, Van Loo P, Dive C, Lin CJ, Rabinowitz M, Aerts HJWL, Hackshaw A, Shaw JA, Zimmermann BG; TRACERx consortium; PEACE consortium; Swanton C. Phylogenetic ctDNA analysis depicts early-stage lung cancer evolution. Nature. 2017 Apr 26;545(7655):446-451. doi: 10.1038/nature22364. PMID 28445469
- [Background] Chaudhuri AA, Chabon JJ, Lovejoy AF, Newman AM, Stehr H, Azad TD, Khodadoust MS, Esfahani MS, Liu CL, Zhou L, Scherer F, Kurtz DM, Say C, Carter JN, Merriott DJ, Dudley JC, Binkley MS, Modlin L, Padda SK, Gensheimer MF, West RB, Shrager JB, Neal JW, Wakelee HA, Loo BW Jr, Alizadeh AA, Diehn M. Early Detection of Molecular Residual Disease in Localized Lung Cancer by Circulating Tumor DNA Profiling. Cancer Discov. 2017 Dec;7(12):1394-1403. doi: 10.1158/2159-8290.CD-17-0716. Epub 2017 Sep 24. PMID 28899864
- [Background] Chen K, Zhao H, Shi Y, Yang F, Wang LT, Kang G, Nie Y, Wang J. Perioperative Dynamic Changes in Circulating Tumor DNA in Patients with Lung Cancer (DYNAMIC). Clin Cancer Res. 2019 Dec 1;25(23):7058-7067. doi: 10.1158/1078-0432.CCR-19-1213. Epub 2019 Aug 22. PMID 31439586
- [Background] Travis WD, Brambilla E, Nicholson AG, Yatabe Y, Austin JHM, Beasley MB, Chirieac LR, Dacic S, Duhig E, Flieder DB, Geisinger K, Hirsch FR, Ishikawa Y, Kerr KM, Noguchi M, Pelosi G, Powell CA, Tsao MS, Wistuba I; WHO Panel. The 2015 World Health Organization Classification of Lung Tumors: Impact of Genetic, Clinical and Radiologic Advances Since the 2004 Classification. J Thorac Oncol. 2015 Sep;10(9):1243-1260. doi: 10.1097/JTO.0000000000000630. PMID 26291008
- [Background] Abbosh C, Birkbak NJ, Swanton C. Early stage NSCLC - challenges to implementing ctDNA-based screening and MRD detection. Nat Rev Clin Oncol. 2018 Sep;15(9):577-586. doi: 10.1038/s41571-018-0058-3. PMID 29968853
- [Derived] Yang H, Gu X, Wang Z, Liu G, Niu Y, Pan X, Yao F. Predicting non-small cell lung cancer lymph node metastasis: integrating ctDNA mutation/methylation profiling with positron emission tomography-computed tomography (PET-CT) scan: protocol for a prospective clinical trial (LUNon-invasive Study). J Thorac Dis. 2024 Sep 30;16(9):6272-6285. doi: 10.21037/jtd-24-1033. Epub 2024 Sep 26. PMID 39444874